CLINICAL TRIAL: NCT06770127
Title: Efficacy of La Roche Posay Routine in the Management of Facial Post Inflammatory Hyperpigmentation (PIHP)
Acronym: PIHP
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP 22048-Serum
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2023-10

CONDITIONS: Acne; Postinflammatory Hyperpigmentation
MeSH Terms: conditions — Acne Vulgaris; Hyperpigmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Routine La Roche Posay: Niacinamide A serum and UV Mune
- Routine Thiamidol: Eucerin Thiamidol antipigment serum and Eucerin SPF50+

SUMMARY:
The goal of this clinical trial is to test and compare La Roche Posay routine --the studied product-- with a comparator product in participants with acne. The main question it aims to answer is how well can the product de-pigment the skin.

The participants will be asked to use the products given twice daily. Researchers will compare the routine La Roche Posay group(experimental) with the routine Eucine group(control) to see if the La Roche product shows superiority in case of better efficacy.

DETAILED DESCRIPTION:
The sample size of this study is 80 participants; 40 subjects testing Niacinamide A serum and UV Mune and 40 subjects testing Eucerin Thiamidol anti-pigment serum and Eucerin SPF 50+. The secondary objectives are:

* the effect on the cutaneous acceptability by clinical examination under dermatological control
* the effect of the product on acne lesions is assessed by comparing the number of elements on the face before application and after product use
* the effect on acne severity according to the Global Acne Evaluation
* the mean darkness of the post-inflammatory hyper-pigmentation (PIHP) lesions. A statistical analysis of the following will be done: a comparison of the before/after application, a comparison of the values obtained from the comparison product/comparator product, and a comparison PIHP lesion/normal zone.

The study endpoints are:

* global acne evaluation scale
* mean size, intensity, number of PIHP lesion
* mean darkness of lesions
* subject global assessment score
* improvement in scores in a stigmatization questionnaire
* satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin phototype: III to VI;
* Moderate to severe PIHP due to acne (score PAHPI > 10);
* Subjects with mild acne on the face (GEA = 2);
* ≤ 4 inflammatory lesions total (non-inflammatory lesions could be 0)

Exclusion Criteria:

* Subjects with symptoms of COVID-19 (moderate fever, dry cough and other symptoms described by the World Health Organization);
* Subjects with a temperature above 37.5 °C;
* COVID-19 positive patients;
* For women: pregnant or nursing woman or woman planning to get pregnant during the study;
* Cutaneous pathology on the study zone (eczema, etc);
* Use of topical or systemic treatment (for ex: treatment of acne) during the previous weeks liable to interfere with the assessment of the cutaneous acceptability/efficacy of the study product;
* Subject with make-up products on the day of the visit at the laboratory;
* Acne and depigmenting treatment (topical or systemic):
* Topical treatment claiming depigmenting effect of the face: within the last month,
* Facial procedures: within the last 3 months,
* Systemic retinoid: within the last 6 months.
* Cosmetic product for non-comedogenicity within the last 2 weeks;
* Subjects treated for PIHP within the past 3 months with either a cosmetic product or a drug;
* Any change in hormonal treatment (including contraceptive) during the three previous months of the study;
* Subject having undergone a surgery under general anesthesia within the previous month;
* Excessive exposure to sunlight or UV-rays within the previous month;
* Subject enrolled in another clinical trial during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with Fitzpatrick skin phototype III to VI who have moderate to severe PIHP due to acne (score PAHPI >10). Subjects with mild face acne (GEA = 2) and ≤4 total inflammatory lesions (including 0).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Clinical scoring of the post-acne hyperpigmentation index | 84 days
  The scoring performed by the investigator on day 0, day 28, day 56 and day 84 from the day of product use. Descriptive statistics where the frequency and percentage frequency of mean size, intensity, number of PIHP lesions and the global score will be calculated to infer the effect of the product on the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Randamy, Study Director — Insight Research
Locations (1):
- Insight Research, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No